CLINICAL TRIAL: NCT02816177
Title: Impact of Telemedicine on Avoiding Emergency Hospital Admissions and Hospitalization for Nursing Home Residents
Brief Title: Telemedicine and Nursing Home
Acronym: GERONTACCESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: I14036/GERONTACCESS
Record Dates: First submitted 2016-06-24; First posted 2016-06-28 (Estimated); Last update posted 2025-07-16 (Actual); Status verified 2019-01

CONDITIONS: Elderly; Multimorbidity
MeSH Terms: interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telemedicine (Experimental): Usual care and telemedicine consultations during12 months.
  Interventions: Other: Telemedicine; Other: Usual Care
- Usual care alone (Active Comparator): Usual care during12 months.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Telemedicine
  Arms: Telemedicine
Other: Usual Care

SUMMARY:
Telemedicine-based care provides remote health and social care to maintain people's autonomy and increase their quality of life. The rapidly aging population has come with a significant increase in the prevalence of chronic diseases and their effects, and thus the need for increased care and welfare.

This solutions give a new opportunity for diagnosis, treatment, education, and rehabilitation, and make it possible to monitor patients with a number of chronic diseases. It also reduces socioeconomic disparity with regard to access to care and gives equal chances to patients from urban and rural areas.

This a randomized trial of telemedicine versus usual care alone to reduce hospitalization and emergency hospital admissions for Nursing Home Residents .

After an initial assessment , each participant is monitored by teleconsultation on six occasions over 12 months. Patients with usual care have an initial and a 12 months assessments.

ELIGIBILITY:
Inclusion Criteria:

* Elderly over 60 years

  * Resident in nursing homes
  * Resident with multiples chronic diseases with at least two comorbidities
  * Having given free and informed consent in writing and signed by himself and / or his legal representative

Exclusion Criteria:

* Resident unaffiliated or not beneficiary of Social Security
* Resident with a life-threatening disease

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 428 (Actual)
Dates: Start 2016-07-05 (Actual); Primary Completion 2018-01-18 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Efficacy | 12 month
  Proportion of patients who had an admission to the emergency or unscheduled hospitalization in health service or surgery

SECONDARY OUTCOMES:
MAST | 12 months
  Cost / effectiveness of telemedicine based on the MAST model (Model of Assessment of Telemedicine ).

CONTACTS AND LOCATIONS:
Overall Officials: Thierry DANTOINE, MD, Principal Investigator — CHU Limoges
Locations (1):
- Service de Gériatrie, Limoges, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Gayot C, Laubarie-Mouret C, Zarca K, Mimouni M, Cardinaud N, Luce S, Tovena I, Durand-Zaleski I, Laroche ML, Preux PM, Tchalla A. Effectiveness and cost-effectiveness of a telemedicine programme for preventing unplanned hospitalisations of older adults living in nursing homes: the GERONTACCESS cluster randomized clinical trial. BMC Geriatr. 2022 Dec 22;22(1):991. doi: 10.1186/s12877-022-03575-6. PMID 36550496